CLINICAL TRIAL: NCT05618236
Title: Comparison of Sugammadex and Neostigmine in Terms of Awakening, Pain, Agitation, Nausea and Vomiting in Pediatric Patients''
Brief Title: Sugammadex and Neostigmine in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Meliha Orhon, assistant professor, Marmara University
Other Study IDs: 09.2022.98
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Vomiting; Postoperative Nausea; Postoperative Delirium
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Emergence Delirium | interventions — Sugammadex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neostigmin+atropin: This will be the group of patients decurarized with neostigmine+atropine,
  Interventions: Drug: Group N; neostigmine+atropine
- sugammadeks: This will be the group of patients decurarized with sugammadex.
  Interventions: Drug: GROUP S; decurarized with sugammadex.

INTERVENTIONS:
Drug: Group N; neostigmine+atropine — The patients included in the study will be divided into 2 groups according to the agent used in decurarization. There is no condition for the number of patients in the group to be equal. Group N; neostigmine+atropine, GROUP S; This will be the group of patients decurarized with sugammadex.
  0-45 days after patients are extubated. And at the 2nd hour, FLACC Scale (Pain Diagnostic Scale), PAED (Pediatric Anesthesia Recovery Delirium) Scale assessment methods will be compared in terms of pain and agitation. Nausea and vomiting will be noted as yes/no.
  Other Names: neostigmine+atropine
  Groups: neostigmin+atropin
Drug: GROUP S; decurarized with sugammadex. — The patients included in the study will be divided into 2 groups according to the agent used in decurarization. There is no condition for the number of patients in the group to be equal. Group N; neostigmine+atropine, GROUP S; This will be the group of patients decurarized with sugammadex.
  0-45 days after patients are extubated. And at the 2nd hour, FLACC Scale (Pain Diagnostic Scale), PAED (Pediatric Anesthesia Recovery Delirium) Scale assessment methods will be compared in terms of pain and agitation. Nausea and vomiting will be noted as yes/no.
  Other Names: sugammadex
  Groups: sugammadeks

SUMMARY:
In this study, it was aimed to compare the use of sugammadex instead of neostigmine + atropine in the reversal of NMB in children undergoing lower abdominal surgery or urogenital surgery, and to compare the rates of postoperative agitation, nausea and vomiting using the FLACC scale, PAED scale and ICC parameters.After the approval of the local ethics committee and written consent from the family, patients who underwent ASA 1, 5-12 years old lower abdomen surgery or urogenital surgery in Pendik Training and Research Hospital will be included in the study.

The patients included in the study will be those who were maintained with routine 2-3% sevoflurane inhalation anesthetic and 0.2mcg/kg/min remifentanil intravenous anesthetic, and decurarized with 0.5-1 mg/kg rocuronium. No drugs other than those administered by the responsible Anesthesiologist during the operation will be administered.

The patients included in the study will be divided into 2 groups according to the agent used in decurarization. There is no condition for the number of patients in the group to be equal. Group N; neostigmine+atropine, GROUP S; This will be the group of patients decurarized with sugammadex.

0-45 days after patients are extubated. And at the 2nd hour, FLACC Scale (Pain Diagnostic Scale), PAED (Pediatric Anesthesia Recovery Delirium) Scale assessment methods will be compared in terms of pain and agitation. Nausea and vomiting will be noted as yes/no.

DETAILED DESCRIPTION:
Lower abdominal surgery and urogenital surgery are frequently performed surgeries in the pediatric patient population aged 5-12 years. Therefore, pain, agitation, nausea and vomiting occurring in the early postoperative period and afterwards are important problems for pediatric patients. The incidence of agitation, which is a postoperative behavioral disorder due to the use of sevoflurane and desflurane, varies between 2 and 80%, depending on the scoring system and anesthesia technique. It is more common in preschool children (3-5 years). Agitation despite spontaneous resolution; It is still considered a potentially serious complication due to the risks of self-harm and the stress it causes in the family. It can also cause pain and bleeding, prolonging the recovery period (1). Therefore, it is a problem that should be avoided.

Neostigmine is the most commonly used agent for reversing neuromuscular blockade (NMB) (2). Cholinesterase inhibitor agents used in decurarization have serious side effects, especially because they stimulate the muscarinic system as well as nicotinic receptors (3). These are hypersalivation, bradycardia, bronchoconstriction, nausea and vomiting, and abdominal cramps (4).

Sugammadex is a cyclodextrin group drug, which is an aminosteroid neuromuscular blocking agent, has a selective effect on rocuronium and vecuronium and mechanically binds these molecules, providing rapid excretion and decurarization. Recurarization and muscarinic side effects are not expected in this type of decurarization(5). When acetylcholine esterase inhibitors are used to reverse neuromuscular block, they can cause postoperative residual curarization (PORC)(6).

Postoperative nausea and vomiting (PONV) is a common complication in the pediatric population. The incidence in children varies between 33.2% and 82% depending on the risk factors of the patient. This rate is twice that of adults. PONV typically describes nausea, vomiting, or retching. It may start in the recovery unit and continue for 24 hours. PONV causes dehydration, electrolyte disturbances, longer stay in the recovery unit, A< it causes delays and ultimately a significant financial burden(7). Therefore, it is a complication that should be avoided as much as possible.

Pain is the most important risk factor in the development of agitation. In order to reduce all these complications, we hypothesized that sugammadex was superior to neostigmine + atropine in reducing side effects compared to decurarization.In this study, it was aimed to compare the use of sugammadex instead of neostigmine + atropine in the reversal of NMB in children undergoing lower abdominal surgery or urogenital surgery, and to compare the rates of postoperative agitation, nausea and vomiting using the FLACC scale, PAED scale and ICC parameters.After the approval of the local ethics committee and written consent from the family, patients who underwent ASA 1, 5-12 years old lower abdomen surgery or urogenital surgery in Pendik Training and Research Hospital will be included in the study.

The patients included in the study will be those who were maintained with routine 2-3% sevoflurane inhalation anesthetic and 0.2mcg/kg/min remifentanil intravenous anesthetic, and decurarized with 0.5-1 mg/kg rocuronium. No drugs other than those administered by the responsible Anesthesiologist during the operation will be administered.

The patients included in the study will be divided into 2 groups according to the agent used in decurarization. There is no condition for the number of patients in the group to be equal. Group N; neostigmine+atropine, GROUP S; This will be the group of patients decurarized with sugammadex.

0-45 days after patients are extubated. And at the 2nd hour, FLACC Scale (Pain Diagnostic Scale), PAED (Pediatric Anesthesia Recovery Delirium) Scale assessment methods will be compared in terms of pain and agitation. Nausea and vomiting will be noted as SPSS 22.0 program will be used in statistical analysis. Mean, standard deviation, median lowest, highest, frequency and ratio values will be used in the descriptive statistics of the data. The distribution of variables will be measured with the Kolmogorov-Smirnov test. Independent sample t-test and mann-whitney u-test will be used in the analysis of quantitative independent data. Paired sample t-test will be used in the analysis of dependent quantitative data. The MC Nemar test will be used in the analysis of dependent qualitative data. Repeated Measure Anova will be used in the analysis of repeated measurements. The fischer test will be used when the conditions for the -square test and chi-square test in the analysis of qualitative independent data are not met.

Power analysis was performed using the G*Power (v3.1.7) program to determine the number of samples. The power of the study is expressed as 1-β (β = probability of Type II error) and in general studies should have 80% power. According to Cohen's effect size coefficients; According to the calculation made by assuming that the evaluations to be made between two independent groups will have a medium effect size (d=0.50), there must be at least 65 people in the groups to achieve 80% power at the α=0.05 level.

ELIGIBILITY:
Inclusion Criteria:

After the approval of the local ethics committee and written consent from the family ASA 1 5-12 years old

Exclusion Criteria:

history of allergy or anaphylaxis to one of the drugs used children with autism children with auditory problems family without consent

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: ASA 1, patients aged 5-12 years who will undergo lower abdominal surgery or urogenital surgery
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
postoperative delirium | postoperatif first 2 hours.
  after patients are extubated. Evaluation Pediatric Anesthesia Recovery Delirium Scale at 2nd Hour

SECONDARY OUTCOMES:
postoperative pain | postoperatif first 2 hours.
  after patients are extubated. Evaluation of Pain Diagnostic Scale

CONTACTS AND LOCATIONS:
Overall Officials: MELIHA ORHON ERGUN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)